CLINICAL TRIAL: NCT06090474
Title: An Open-label, One-sequence, Three-period, Multiple-dose Study to Evaluate Drug-drug Interactions, Safety and Tolerability Between NDC-002A/NDC-002B and NDC-002C in Healthy Volunteers
Brief Title: Multiple Dose Study to Evaluate Drug-drug Interactions, Safety and Tolerability of NDC-002 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Noah Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NDC002-P001
Record Dates: First submitted 2023-10-06; First posted 2023-10-19 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Stroke Sequelae; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NDC-002 (Experimental): In Period 1, Two tablets of NDC-002C are repeatedly administered once a day for seven days to reach a steady state of NDC-002C. There is a seven-day washout period between Period 1 and Period 2.
  In Period 2, after repeated administration of one tablet of NDC-002A once a day for seven days, one tablet of NDC-002B is administered repeatedly once a day for eight days to reach a steady state of NDC-002B.
  In Period 3, after the completion of Period 2 administration and without a washout period, one tablet of NDC-002B and two tablets of NDC-002C administered repeatedly in combination once a day for seven days.
  Interventions: Drug: NDC-002

INTERVENTIONS:
Drug: NDC-002 — Combination of NDC-002B and NDC-002C

SUMMARY:
An Open-label, One-sequence, Three-period, Multiple-dose Study to Evaluate Drug-drug Interactions, Safety and Tolerability between NDC-002A/NDC-002B and NDC-002C in Healthy Volunteers

DETAILED DESCRIPTION:
This is an Open-label, One-sequence, Three-period, Multiple-dose Study and the goal of this clinical trial is to evaluate in health Volunteers.

The main question[s] it aims to answer are:

* Drug-drug Interactions
* Safety
* Tolerability

The study consisted of Three-period: Period 1 which repeated administration of NDC-002C for 7 days and Period 2 which repeated administration of NDC-002A for 7 days, followed by administration of NDC-002B for 8 days and Period 3 which repeated concomitant administration of NDC-002B and NDC-002C for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged between 19 and 55 at the time of screening
2. For men, those who weigh 50 kilograms or more and for women, those who weigh 45 kilograms or more and have a body mass index (BMI) between 18.0 and 30.0
3. Those who do not have any congenital or chronic disease and had no pathological symptoms or findings in a medical examination
4. Those who are deemed suitable as subjects by the investigator within four weeks prior to the first administration date of the investigational product based on the characteristics of the drug as a result of interview, physical examination, clinical laboratory test, and electrocardiogram
5. Those who are able to understand and follow instructions and participate throughout the entire clinical trial period
6. Those who agree to contraception use during the clinical trial period and can comply with medically accepted contraceptive methods (including those who are medically infertile)
7. Those who have heard and fully understood a detailed description of this clinical trial and have voluntarily decided to participate in the trial and have agreed in writing to comply with the precautions

Exclusion Criteria:

1. Medical History

   1. Those with or with a history of clinically significant diseases of the biliary system (biliary obstructive disease, etc.), renal system (severe renal failure, etc.), blood/oncology, cardiovascular system (congestive heart failure, coronary or aortic/mitral stenosis or complications thereof, arrhythmia, renovascular hypertension, etc.), respiratory system (asthma, chronic obstructive pulmonary disease, etc.), liver (moderate or severe liver failure, etc.), endocrine system (diabetes or impaired glucose tolerance, hypothyroidism, primary aldosteronism, etc.), digestive system, musculoskeletal system, or central nervous system disease (Parkinson's disease, etc.), or mental illness or malignant tumor
   2. Those with a history of gastrointestinal disease (Crohn's disease, ulcers, gastritis, gastrospasms, gastroesophageal reflux, acute or chronic pancreatitis, etc.) or gastrointestinal surgery (except simple appendectomy or hernia surgery) that may affect drug absorption
   3. Those with a history of hypersensitivity or clinically significant hypersensitivity to donepezil or drugs containing NAC or similar agents (piperidine derivatives, etc.), or other drugs (aspirin, antibiotics, etc.)
   4. Those who have suffered from a clinically significant disease within 30 days before the first administration of the investigational product
2. Clinical Laboratory Tests

   1. Those with systolic blood pressure ≥ 140 mmHg or ≤ 99 mmHg, or diastolic blood pressure ≥ 91 mmHg or ≤ 59 mmHg, or measured pulse rate ≥ 101 or ≤ 40 times per minute for vital signs measured in a sitting position after sufficient rest
   2. Those who are tested positive for serological tests (hepatitis B, hepatitis C, syphilis, HIV)
   3. Patients with active liver disease, including a persistent increase of liver enzyme levels (AST, ALT) of unknown etiology or an increase of liver enzyme levels ≥ 1.5 times the ULN
   4. Patients with renal impairment of moderate or higher renal failure (GFR <60 mL/min based on the Cockcroft-Gault method)
   5. Patients with CPK values increased by more than five times the ULN
   6. In the case of clinically significant findings on an electrocardiogram or related physical abnormalities or symptoms
   7. If the investigator determines that it is difficult to proceed with the trial due to results of physical examinations
3. Allergies and Drug Abuse

   1. Those with genetic problems such as intolerance to the additivies for donepezil or NAC
   2. Those with a history of drug abuse or who tested positive for drug abuse in the drug screening test
   3. Those with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
4. Contraindicated Concomitant Drugs/Diet

   1. Those who have participated in other clinical trials within 180 days before the first administration of the investigational product
   2. Those who have taken metabolism-inducing or inhibiting drugs (CYP2D6 or CYP3A4 inducers, inhibitors, etc.) within 28 days before the first administration of the investigational product
   3. Those who have taken herbal medicine within 28 days, prescription drugs within 14 days, or over-the-counter drugs within seven days before the first administration of the investigational product (however, if other conditions are reasonable, at the discretion of the investigator, the subject may participate in the clinical trial)
5. Other

   1. Those who have done whole blood donation within 60 days, or apheresis within 28 days before the first administration of the investigational product, or received a blood transfusion within 28 days before the first administration
   2. Those who have consumed excessive alcohol within 28 days before the first administration (alcohol > 30 g/day; soju > 150 cc/day (based on 20%), beer > 750 cc/day (based on 4%), liquor > 75 cc/day (based on 40%) , wine > 300 cc/day (based on 10%))
   3. Those who have smoked excessively within 28 days before the first administration (cigarettes > 10 cigarettes/day) or those who could not quit smoking during the clinical trial
   4. Those who have consumed excessive caffeine within 28 days before the first administration (coffee > 5 cups/day, tea > 1250 cc/day, coke 1250 cc/day)
   5. Those who consume alcohol continuously or are unable to abstain from alcohol during the clinical trial
   6. Those who are judged unsuitable for participation in the clinical trial by the investigator (study doctor) for other reasons, including the results of clinical laboratory tests

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Safety Evaluation: Adverse events | Up to 10 days post final dose
  Subjective/objective symptoms
Pharmacokinetic Evaluation: AUCss,τ of NDC-002B/C | Day 1, Day 7, Day15, Day 29, Day 36
  after single and concomitant administration of NDC-002B/C
Pharmacokinetic Evaluation: Css,max of NDC-002B/C | Day 1, Day 7, Day15, Day 29, Day 36
  after single and concomitant administration of NDC-002B/C

SECONDARY OUTCOMES:
Pharmacokinetic Evaluation: AUCss,inf of NDC-002B/C | Day 1, Day 7, Day15, Day 29, Day 36
  after single and concomitant administration of NDC-002B/C
Pharmacokinetic Evaluation: Tss,max of NDC-002B/C | Day 1, Day 7, Day15, Day 29, Day 36
  after single and concomitant administration of NDC-002B/C
Pharmacokinetic Evaluation: Tss,1/2 of NDC-002B/C | Day 1, Day 7, Day15, Day 29, Day 36
  after single and concomitant administration of NDC-002B/C

CONTACTS AND LOCATIONS:
Locations (1):
- Insan Medical Foundation Metro Hospital, Anyang-si, South Korea

IPD SHARING:
Plan to Share IPD: No